CLINICAL TRIAL: NCT07232394
Title: The Impact of Early Feeding and Mobilization on Rehabilitation in Thoracic Surgery: A Prospective Randomized Controlled Trial
Brief Title: Early Feeding and Mobilization in Thoracic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jianxing He (Other)
Responsible Party: Sponsor-Investigator, Jianxing He, Professor, The First Affiliated Hospital of Guangzhou Medical University
Organization: The First Affiliated Hospital of Guangzhou Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ERAS-VATS01
Record Dates: First submitted 2025-11-13; First posted 2025-11-18 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Thoracic Surgery Lung; Nursing Cares; ERAS
Keywords: ERAS; lung cancer; video-assisted thoracoscopic surgery; nursing care
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ERAS nursing group (Experimental): The ERAS nursing group implements the Enhanced Recovery After Surgery (ERAS) protocol, where the medical team uses developed assessment tools to individualize the timing for each patient's first mobilization and oral intake after surgery. This intervention aims to promote postoperative recovery, reduce postoperative complications, and shorten hospital stays.
  Interventions: Behavioral: Traditional nursing; Behavioral: ERAS protocol
- Traditional nursing group (Active Comparator): The traditional nursing group receives standard postoperative care, including routine nursing interventions for pain management, mobility, and nutrition.
  Interventions: Behavioral: Traditional nursing

INTERVENTIONS:
Behavioral: Traditional nursing — After the patient is admitted, the nursing team conducts a comprehensive assessment, including blood glucose, blood pressure, medication history, smoking history, alcohol consumption history, etc., to develop the patient's care plan. Preoperatively, the nursing staff will educate the patient about perioperative knowledge and inform the patient about fasting and withholding fluids 8 hours before the surgery. Postoperatively, the nursing staff closely monitors the patient's vital signs, surgical wounds, and drainage, and provides relevant health education. According to medical orders, the nursing team will guide the patient in appropriate eating and activity, and use medications to address postoperative discomfort.
Behavioral: ERAS protocol — At 0, 2, and 4 hours postoperatively, the nursing team will progressively assess the patient's condition in the order of vital signs, consciousness, nausea and vomiting severity, swallowing function, pain score, and muscle strength. If all the assessment results meet the criteria, the nursing staff will guide the patient to try eating a small amount of liquid food and maintain the head of the bed elevated to a 30-degree angle. At the same time, the nursing staff will guide the patient to follow a progressive activity regimen, starting with sitting up in bed for 3 minutes, then sitting at the bedside for 3 minutes, followed by standing at the bedside for 3 minutes. If there is no discomfort, the patient may walk moderately within the ward.
  Arms: ERAS nursing group

SUMMARY:
This study evaluates the safety and effectiveness of an innovative care assessment tool for early feeding and mobilization following thoracic surgery, based on the Enhanced Recovery After Surgery (ERAS) protocol. The aim is to improve postoperative recovery by helping healthcare providers implement a structured, evidence-based plan for early feeding and activity. The study will compare the new care model (ERAS-based) with traditional postoperative care. The investigators will focus on outcomes like recovery quality, complications, hospital stay, and medication use. This research aims to provide solid evidence for integrating early feeding and mobilization into routine thoracic surgery recovery, potentially improving patient comfort, reducing recovery time, and lowering complications.

DETAILED DESCRIPTION:
Lung cancer remains the leading cause of cancer-related morbidity and mortality worldwide. Surgery, especially for early and intermediate-stage patients, is considered the cornerstone of treatment. With the advancement of minimally invasive techniques, such as video-assisted thoracic surgery (VATS), the degree of surgical trauma and the risk of complications have significantly decreased. However, despite these innovations, postoperative complications still occur in 30%-40% of patients, indicating that improvements in surgical techniques alone are insufficient to eliminate perioperative risks.

In response, the Enhanced Recovery After Surgery (ERAS) protocol has been introduced in thoracic surgery to optimize postoperative recovery. ERAS strategies have shown promising results in reducing complications, pain medication use, and hospital stays. However, most of the clinical evidence supporting ERAS comes from colorectal surgery, with limited research focusing on its application in thoracic surgery. Further validation of its safety, feasibility, and effectiveness in thoracic surgery patients is urgently needed.

One core element of ERAS in thoracic surgery is early postoperative oral feeding. Traditional postoperative management often restricts food and fluids for 4-6 hours to reduce the risk of nausea and vomiting caused by residual anesthesia, but this restriction can lead to discomfort from thirst and hunger. Restoring oral intake as early as possible, provided there is no high aspiration risk and vital signs are stable, has been shown to enhance comfort and recovery. However, clinical implementation of early feeding has been suboptimal, and most related studies have focused on gastrointestinal surgeries. Evidence supporting early feeding in thoracic surgery is still lacking.

In addition to early feeding, early mobilization is another key component of ERAS in thoracic surgery. As the ERAS concept evolves, research has increasingly focused on multi-faceted interventions, suggesting that combining early feeding and mobilization could have a synergistic effect in optimizing postoperative outcomes. Despite this potential, high-quality evidence supporting this combined strategy in thoracic surgery is still limited.

Given these challenges, this study aims to evaluate the safety and effectiveness of a newly developed, time-point-based nursing assessment tool for early feeding and mobilization after thoracic surgery. This single-center, randomized, single-blind, parallel-controlled trial will assess the tool's impact on patient outcomes, including recovery quality, complications, and hospital stay. The ultimate goal is to provide evidence for the clinical adoption and implementation of this tool in thoracic surgery recovery, enhancing patient recovery and contributing to the broader application of ERAS principles in this field.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 to 75 years, with no gender restrictions;
2. Planned for elective thoracoscopic surgery, in good physical condition, able to undergo surgery and anesthesia (ASA classification no more than class III), and confirmed suitable for surgery after joint assessment by the medical and nursing team;
3. No severe cognitive impairment or mental illness, able to cooperate with nursing staff and follow intervention measures;
4. Normal function of major organs;
5. The patient has provided informed consent to participate in the study and signed the informed consent form.

Exclusion Criteria:

1. Patients with cognitive impairment, mental illness, or other conditions that may affect the study;
2. Requirement to convert to open surgery during the procedure;
3. Lung cancer with metastasis to other organs;
4. Failure to sign the informed consent form.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 232 (Actual)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2025-09-01 (Actual)

PRIMARY OUTCOMES:
The Quality of Recovery-15 (QoR-15) score | 24 hours post-surgery.
  The QoR-15 scale is a 15-item questionnaire used to assess the patient's quality of life during the postoperative recovery process, covering aspects such as pain, fatigue, anxiety, physical function, and emotional recovery. The higher the total score, the better the postoperative recovery quality.

SECONDARY OUTCOMES:
Chest Tube Placement Duration | Perioperative.
  The chest tube placement duration refers to the number of days from the placement of the chest tube after surgery until its removal.
Total Drainage Volume from Chest Tube | Perioperative.
  The total drainage volume from the chest tube refers to the total amount of fluid drained through the chest tube after surgery.
Postoperative Hospitalization Duration | Perioperative.
  The postoperative hospitalization duration refers to the total number of days the patient remains in the hospital from the completion of surgery until discharge.
Postoperative Complications | Perioperative.
  Postoperative complications refer to any adverse events or symptoms that occur after surgery and may affect the patient's recovery.
Total Hospitalization Costs | Perioperative.
  The total cost of hospitalization includes all medical expenses, such as surgical fees, inpatient care, medication costs, and examination fees.
30-Day Readmission Rate | Within 30 days post-surgery.
  The proportion of patients readmitted to the hospital within 30 days after surgery for any reason.
30-Day Mortality Rate | Within 30 days post-surgery.
  The mortality rate within 30 days after surgery due to any cause.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No